CLINICAL TRIAL: NCT05181098
Title: Prospective Robotic-Guided Registry of Spine Surgery
Acronym: PRoGRSS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The National Spine Health Foundation (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: ROB-002
Record Dates: First submitted 2021-09-10; First posted 2022-01-06 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Spinal Disease
Keywords: Robotic-guided spine surgery
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Robotic-guided surgery group: Any pediatric, adolescent or adult patient undergoing robotic-guided spine surgery, ages 12-80.
  Interventions: Procedure: Robotic-guided spine surgery

INTERVENTIONS:
Procedure: Robotic-guided spine surgery — The Mazor X Stealth Edition robotic platform will be used to guide posterior instrumentation during spine fusion surgery.

SUMMARY:
This study aims to combine multi-center data of robotic assisted spine surgery, to evaluate the true scope of this advancing technology.

DETAILED DESCRIPTION:
What is the impact on clinical and patient-reported outcomes for participants who undergo robot assisted surgery? This will be the first multi-center study to prospectively collect data on robotic assisted spine surgery outcomes. The primary objective of this study will be to facilitate quantification of potential short- and long-term benefits of robotically guided spine surgeries.

It is hypothesized that use of robotic guidance during spinal instrumentation will have numerous short- and long-term benefits to both participant and surgeon. Expected benefits include improved surgical and clinical outcomes, lower incidence of procedure-related adverse events (e.g., fewer new neurological deficits, implant-related durotomies, and implant misplacements), improved implant accuracy, lower intraoperative radiation exposure, and lower reoperation rates, when compared to the published literature.

The secondary objective of this study is to assess the clinical performance of robotic instrumentation as per the pre-operative plan. To this end, data on a number of common clinical metrics will be analyzed to determine the extent to which they are affected by the use of robotic guidance during implantation.

ELIGIBILITY:
Inclusion Criteria:

* Any pediatric, adolescent or adult patient
* Undergoing open or MIS robotic-guided spine surgery using the Mazor Core Technology.

Exclusion Criteria:

* Pregnancy
* active infection
* malignancy
* primary abnormalities of bone
* primary muscle diseases (e.g., muscular dystrophy)
* neurologic diseases
* spinal cord abnormalities/lesions
* paraplegia.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any pediatric, adolescent or adult patient undergoing robotic-guided spine surgery, ages 12-80.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the success of robotic-guided spine surgery, from planning to execution. | 1 year after surgery
  To evaluate the success from planning to execution of robotic screw placement.
To evaluate the success of robotic-guided spine surgery, by screw placement accuracy. | 1 year after surgery
  To determine screw accuracy
To evaluate the success of robotic-guided spine surgery, by revision surgery rates. | 1 year after surgery
  To determine the rate of revision surgery due to symptomatic screw malposition within 1 year
To evaluate the success of robotic-guided spine surgery, by the radiation exposure. | 1 year after surgery
  To determine radiation exposure to the patient and surgeon.

SECONDARY OUTCOMES:
To evaluate clinical outcomes, as determined by all cause revisions | 1 year after surgery
  To determine the rate of revision surgery for all causes within 1 year
To evaluate clinical outcomes, by surgical complications | 1 year after surgery
  To determine the rate of surgical complications (wound infection/dehiscence, major neurological deficit, hemorrhage, dural tear)
To evaluate clinical outcomes, by patient reported outcome measures | 1 year after surgery
  To evaluate for changes in Patient Reported Outcomes Measurement Information System (PROMIS) scores over 1 year; (PROMIS scores are calculated at T-scores on a 0-100 point scale - for positively worded functions, such as physical function and global health, the higher the score the better the outcome; but for negatively worded functions, like pain interference, the higher the score the worse the outcome).
To evaluate clinical outcomes, by patient disability rating | 1 year after surgery
  To evaluate for changes in Oswestry Disability Index (ODI) scores over 1 year; disability scores range from 0-100, the higher the score the worse the outcome/disability.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Good, MD, Principal Investigator — Virginia Spine Institute
Locations (1):
- National Spine Health Foundation, Reston, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data.